CLINICAL TRIAL: NCT04838054
Title: Pilot Study: The Efficacy of Stabilized Chlorine Dioxide Rinse as a Chemical Adjuvant for Treatment of Peri-implant Mucositis
Brief Title: The Efficacy of Stabilized Chlorine Dioxide Rinse as a Chemical Adjuvant for Treatment of Per-implant Mucositis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rowpar Pharmaceuticals, Inc. (Industry)
Collaborators: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00024706
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Results first posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Intervention Model Description: Subjects will receive an Oral Hygiene Kit at Visit 1. The MGI, BOP and PI, Pocket depth and radiographs will be measured and all oral tissues examined (baseline examination). Subjects will return for Visit 2 in 14 days ± 3 days to: 1) assess and record changes in indices and oral health and any adverse conditions. Visit 3 (45 days ± 7) will be a compliance visit for study drug utilization. Visit 4 (90 days ± 7) will be a repeat of Visit 1.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Once a subject has been screened and qualified for study participation, that subject will be enrolled and assigned the next available randomization number. The study randomization table will be generated by a third-party statistician. This procedure will be used to keep the Study Statistician blinded to subject treatments prior to database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test - stabilized chlorine dioxide rinse (Experimental): Subjects will receive CloSYS Ultra Sensitive Rinse
  Interventions: Drug: Stabilized chlorine dioxide oral rinse
- Placebo - oral rinse, no active ingredients (Placebo Comparator): Subjects will receive oral rinse - no active ingredients
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Stabilized chlorine dioxide oral rinse — Patients received stabilized chlorine dioxide rinse associated with periodontal basic therapy.
  Arms: Test - stabilized chlorine dioxide rinse
Other: Placebo — Patients received a rinse containing no active ingredients and periodontal basic therapy.
  Arms: Placebo - oral rinse, no active ingredients

SUMMARY:
A full understanding of etiology and diagnosis of peri-implant diseases is crucial for finding effective treatments for these diseases that are more widely accessible to dentists. Several treatment protocols for peri-implant diseases have been proposed, but no gold standard has been established to date. Thus, the purpose of this study is to analyze efficacy of stabilized chlorine dioxide as a chemical adjuvant for treatment of peri-implant mucositis in a non-surgical treatment protocol with a 3-month follow-up.

DETAILED DESCRIPTION:
Fifty individuals with peri-implant mucositis will be identified to participate in this study and randomized into two groups to analyze clinical parameters and results of this study: 1) test group (stabilized chlorine dioxide rinse) and 2) control group (placebo). Each group will be associated with periodontal basic therapy.

Treatment Protocol After inclusion of the patients, medical history and initial examination are performed, patients will be randomly divided into the following two groups: 1) test (stabilized chlorine dioxide rinse associated with periodontal basic therapy); and 2) control (placebo associated with periodontal basic therapy).

Periodontal basic therapy will consist of oral hygiene instruction, motivation, retentive factor removal, and an adaptation of the protocol of full-mouth scaling and root planing (stabilized chlorine dioxide mouthwash will be used). Plastic currets are used to instrument the implants and metal currets to instrument teeth. Immediately after instrumentation, chemical solutions of chlorine dioxide or placebo will be dispensed to the subjects.

The subjects will follow their normal oral-hygiene procedures with the addition of using the study rinse toothbrush and toothpaste provided to them.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of peri-implant mucositis
* at least one implant
* probing depth (PD) ≤5mm
* BOP (bleeding on probing)
* No radiographic evidence of bone loss beyond the first two threads of the implant

Exclusion Criteria:

* Active Periodontitis or Peri-implantitis which requires definitive treatment.
* Presence of oral local mechanical factors that could (in the opinion of the PI) influence the outcome of the study.
* Presence of orthodontic appliances, or any removable appliances, that impinges on the tissues being assessed.
* Presence of soft or hard tissue tumors of the oral cavity.
* Patients treated with systemic antibiotic therapy or periodontal/mechanical/local delivery therapy within 12 weeks prior to study entry and throughout the study duration.
* Patients chronically (i.e. two weeks or more) treated with non-steroidal anti-inflammatory drugs (NSAIDs) or any medications know to affect soft tissue condition (excluding treatment of Acetylsalicylic acid ≤ 100 mg/day).
* Patients with uncontrolled diabetes, of any type, and/or patients with HbA1c test value >7.5% dated 3 months prior to the screening visit.
* Patients receiving radiation therapy to the head and neck area and/or receiving immunosuppressive therapy.
* The presence of any medical or psychiatric condition or any other condition that, in the opinion of the Investigator, could affect the successful participation of the patient in the study.
* Drug and alcohol abuse.
* Patient participates in any other clinical study 30 days prior to the start of the study and throughout the study duration.
* Subject is pregnant (based on pregnancy result) or lactating.
* Subject is a smoker, or has been a smoker within the past 6 months.
* Any other condition that may interfere with the study as judged by the PI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas RM Venkatasatya, DDS, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 57 Individuals with peri-implant muscositis were identified to participate in this study and randomized into 2 groups. Each group was associated with periodontal basic therapy.
Pre-assignment Details: No event occurred before participant enrollment.
Period: Overall Study
Arm/Group | Test - Stabilized Chlorine Dioxide Rinse | Placebo - Oral Rinse, no Active Ingredients
Started | 29 | 28
Completed | 27 | 28
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: The focus of the analysis is on the teeth. The study will evaluate the outcome for all teeth as well as compare the outcomes between teeth and implants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test - Stabilized Chlorine Dioxide Rinse | Placebo - Oral Rinse, no Active Ingredients | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 11 | 17
  >=65 years | 23 | 17 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 17 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 26 | 26 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 25 | 22 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Global Probing Depth
Description: The distance measured from the base of the pocket to the most apical point on the gingival margin. Measured in mms. Over 3 mm indicates a need for periodontal therapy. Higher results mean a worse outcome.
Time Frame: 90 days
Population: 29 subjects in the test group and 28 subjects in the placebo group were enrolled. However, 2 subjects from the test group did not complete the study and therefore were excluded from the analysis. So 27 subjects in the test group and 28 placebo subjects were included.
Measure: Mean (Standard Error); unit: mm
Units Other Than Participants: Teeth
Arm/Group | Test - Stabilized Chlorine Dioxide Rinse | Placebo - Oral Rinse, no Active Ingredients
Number analyzed (Participants) | 27 | 28
Number analyzed (Teeth) | 864 | 896
mm | 2.37 (0.166) | 2.64 (0.130)
Statistical Analysis 1: Comparison: Test - Stabilized Chlorine Dioxide Rinse vs Placebo - Oral Rinse, no Active Ingredients; Test type: Superiority; p = 0.28, ANCOVA — p-values <0.05 means statistically significant; Mean Difference (Net) = 0.27

2. Primary Outcome: Global Plaque Score.
Description: The plaque index assesses the amount of dental plaque visible on the vestibular and lingual surfaces of all teeth, except the third molars. The index is calculated by dividing the number of plaque-containing surfaces by the total number of available surfaces. Values range from 0-18 with 0 being excellent and 18 poor. Higher numbers mean a worse outcome.
Time Frame: 90 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Number of Teeth
Arm/Group | Test - Stabilized Chlorine Dioxide Rinse | Placebo - Oral Rinse, no Active Ingredients
Number analyzed (Participants) | 27 | 28
Number analyzed (Number of Teeth) | 864 | 896
score on a scale | 1.57 (0.110) | 1.98 (0.110)
Statistical Analysis 1: Comparison: Test - Stabilized Chlorine Dioxide Rinse vs Placebo - Oral Rinse, no Active Ingredients; Test type: Superiority; p = 0.011, ANCOVA — p<0.05 means statistically significant; Mean Difference (Net) = 0.41

3. Primary Outcome: Modified Gingival Index (MGI)
Description: The MGI relies on a visual assessment of gingival changes to measure the severity of inflammation. Five categories, using a 0-4 scale, score the marginal and papillary gingival tissue based on color, texture, edema, and spontaneous bleeding. 0 being normal and 4 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding. The higher scores mean a worse outcome.
Time Frame: 90 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Number of Teeth
Arm/Group | Test - Stabilized Chlorine Dioxide Rinse | Placebo - Oral Rinse, no Active Ingredients
Number analyzed (Participants) | 27 | 28
Number analyzed (Number of Teeth) | 864 | 896
score on a scale | 1.48 (0.025) | 1.52 (0.035)
Statistical Analysis 1: Comparison: Test - Stabilized Chlorine Dioxide Rinse vs Placebo - Oral Rinse, no Active Ingredients; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 2.99

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Test - Stabilized Chlorine Dioxide Rinse | Placebo - Oral Rinse, no Active Ingredients
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 3/29 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test - Stabilized Chlorine Dioxide Rinse (N=29) | Placebo - Oral Rinse, no Active Ingredients (N=28)
Bitterness in the mouth (Product Issues) | 1 (1) | 0 (0)
Unrelated injury (Social circumstances) | 1 (1) | 0 (0) — Patient sustained knee injury through a fall in the bathroom and was unable to complete the study
Scheduling Issues (Social circumstances) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT04838054/Prot_SAP_000.pdf